CLINICAL TRIAL: NCT04806880
Title: Prospective Study Evaluating the Olfactory Recovery of Anosmia Post COVID-19 by Olfactory Rehabilitation Assisted by Web-application
Brief Title: Study Evaluating the Olfactory Recovery of Anosmia Post COVID-19 by Olfactory Rehabilitation Assisted by Web-application
Acronym: COVIDANOSMIA
Status: Completed | Type: Observational
Sponsor: Weprom (Other)
Collaborators: Kelindi (Industry); Centre National de la Recherche Scientifique, France (Other); Hospital of Tours (Unknown)
Responsible Party: Sponsor
Other Study IDs: WP-2020-06
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: Web-application; Anosmia; COVID-19; coaching
MeSH Terms: conditions — COVID-19; Anosmia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- users: Users of web-application
  Interventions: Device: Web-application

INTERVENTIONS:
Device: Web-application — support for olfactory coaching consisting of the inhalation of fragrant essential oils.

SUMMARY:
Anosmia is a symptom present in 40 to 80% of patients and usually only lasts 1 to 2 weeks. However, in nearly one in five patients, it can last beyond or even several months with consequences in terms of undernutrition and depression. However, olfactory rehabilitation is a technique validated in post-infectious anosmia since 2014 and recommended by international learned societies to accelerate recovery with nearly 63% improvement in anosmia In the context of the health crisis linked to the coronavirus, approximately 1 million French people will have persistent anosmia following an infection with COVID-19. A web-application to support the olfactory coaching of anosmic patients and help with follow-up seems relevant to promote recovery and the proper conduct of this coaching.

covidanosmie.fr is a web application dedicated to olfactory rehabilitation, accessible free of charge.

ELIGIBILITY:
Inclusion Criteria:

* Post-COVID anosmia lasting more than 1 month
* Consent to the use of data via the application

Exclusion Criteria:

* Other causes of anosmia than COVID
* Contraindication to olfactory coaching (allergy to one of the aromatic oils)
* Minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All users of the application who have not objected to the use of their data
Sampling Method: Non-Probability Sample
Enrollment: 1155 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the rate of patients presenting an improvement in their anosmia | 16 weeks
  Number of patients with an improvement in anosmia (increase of at least 1 point on the visual analogue scale 0-10) on the number of users

SECONDARY OUTCOMES:
Evaluation of the time until recovery of at least 1point in 10 (Visual Analog Scale) from anosmia, | 16 weeks
  Time between the date of first use of the application and the date of recovery of at least one point of anosmia
Assessment of the duration of anosmia | 16 weeks
  Time between the date of diagnosis or onset of anosmia and the date of final recovery
Evaluation of the recovery of at least one point in 10 (Visual Analog Scale) depending on the oils | 16 weeks
  Evolution of the VAS according to the different oils, proportion of patients with an increase of at least 1 point in anosmia on a visual analog scale (from 0 no smell to 10 normal smell) of each oil

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice DENIS, MD, Study Director — Weprom
Locations (1):
- ILC, Le Mans, France